CLINICAL TRIAL: NCT01568580
Title: Open-label, Non-comparative, Multicenter, Phase III for Evaluation of Efficacy and Safety of Recombinant Factor VIII (GreenGene) in Previously Treated Patients With Hemophilia A
Brief Title: Efficacy and Safety of Recombinant Factor VIII (GreenGene) in Patients With Hemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC8AIII
Record Dates: First submitted 2012-03-22; First posted 2012-04-02 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Factor VIII; Recombinant
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- test drug (Experimental): GreenGene
  Interventions: Drug: GreenGene

INTERVENTIONS:
Drug: GreenGene — Dose : 10 ~ 50IU/kg Administration method : intravenous infusion or bolus

SUMMARY:
The purpose of this study is to study the evaluation of efficacy and safety of GreenGene (Recombinant Factor VIII).

ELIGIBILITY:
Inclusion Criteria:

* Hemophilia A patients at least 12 years of age
* At least 150 treatment exposure-days to previous FVIII products
* FVIII≤2% at screening or diagnosis (FVIII≤1% for PK study)
* CD4 Lympocyte cell count>400/㎕
* Patients willing to cooperate for the study
* Patient's or legal guardian's consent to participate in the study

Exclusion Criteria:

* FVIII inhibitor(neutralizing antibody to FVIII)≥0.6 Bethesda Units
* Coagulation disorders other than hemophilia A (e.g. Idiopathic Thrombocytopenic Purpura, von Willebrand Disease)
* Platelet count≤100,000㎣
* Subjects with clinical evidence of symptomatic HIV disease regardless of HIV-seroposive/seronegative
* Subjects with rFVIII antibody, mouse IgG antibody, or CHO antibody
* Creatinine levels more than 2 times of reference rage, GOT and GPT levels more than 3 times of reference range, diabetes mellitus or other metabolic disorder
* Subjects with diastolic blood pressure≥100mmHg not controlled with antihypertensive medications
* Anemia(hemoglobin<12g/dL)
* Subjects with severe or life-threatening bleeding just before entry into the trial
* Subjects with a history of treatment failure due to formation of inhibitor to FVIII
* Subjects with a history of severe hypersensitive reactions to FVIII concentrate
* Subjects requiring pre-medication for FVIII infusion(e.g. antihistamines, etc)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2004-12; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Physician's assessment of hemostatic effect for on-demand treatment | 12 months
  Category: Exellent, Good, Moderate, None
Hemostatic effect for major bleeding | up to 1 year
  Category: Exellent, Good, Moderate, None

SECONDARY OUTCOMES:
consumption amount of test drug | up to 12 month or 100 exposure days
Subject's self assessment of treatment | 12 months
  Category: Exellent, Good, Moderate, None
FVIII Recovery(%) | every 3 months
FVIII inhibitor incidence rate | every 3 months
The number of adverse events | up to 1 year
Surgery study: prohylactic effects | up to 1 year
  Category: Exellent, Good, Moderate, None